CLINICAL TRIAL: NCT05057494
Title: A Phase III Prospective, Multicenter, Randomized, Open-Label Trial of Acalabrutinib Plus Venetoclax Versus Venetoclax Plus Obinutuzumab in Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: A Study of Acalabrutinib Plus Venetoclax Versus Venetoclax Plus Obinutuzumab in Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Acronym: MAJIC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8220C00027; 2023-505866-27-00 (Registry Identifier: CTIS); 2021-003936-10 (EudraCT Number)
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Keywords: Chronic lymphocytic leukemia; Small lymphocytic lymphoma; Acalabrutinib; Venetoclax; Obinutuzumab; B-cell lymphoma 2 inhibitors
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Acalabrutinib plus Venetoclax (AV) (Experimental): Participants will receive acalabrutinib and venetoclax orally.
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax
- Arm B: Venetoclax plus Obinutuzumab (VO) (Experimental): Participants will receive Venetoclax orally and Obinutuzumab via IV infusion.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Acalabrutinib — Dose formulation: Capsule or Tablet
  Arms: Arm A: Acalabrutinib plus Venetoclax (AV)
Drug: Venetoclax — Dose formulation: Tablet
Drug: Obinutuzumab — Dose formulation: Injection
  Arms: Arm B: Venetoclax plus Obinutuzumab (VO)

SUMMARY:
A study of acalabrutinib plus venetoclax (AV) versus venetoclax plus obinutuzumab (VO) in previously untreated chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
This is a phase III prospective, multicenter, randomized, open-label trial.

After completion of the screening period, eligible participants will be randomized in a 1:1 ratio to each of the following intervention arms:

Arm A: Minimal Residual Disease (MRD)-limited finite AV therapy Arm B: MRD-limited finite VO therapy

The study consists of screening, treatment, and post-intervention follow-up periods. Participants will undergo safety and efficacy assessments during each period for each study arm. The duration of individual participant involvement in the study will be approximately 5 years.

All participants who discontinue study intervention will be followed for safety assessments and survival status. Safety/survival follow-up is not required if the participant permanently discontinues study intervention due to withdrawal of consent, loss to follow-up, or death

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years at the time of signing the consent form.
2. Documented TN CLL/SLL requiring treatment according to iwCLL guidelines 2018 (Hallek et al 2018).
3. Adequate BM function independent of growth factor or platelet transfusion support within 2 weeks of screening initiation as follows:

   1. Absolute neutrophil count ≥ 1.0 × 10 9 /L; absolute neutrophil count ≥ 500 cells/μL (≥ 0.50 × 109/L) with documented bone marrow (BM) involvement of chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL).
   2. Platelet counts ≥ 30 × 10 9 /L; platelet count ≥ 10 × 10 9 /L in participants with documented BM involvement of CLL/SLL.
4. Estimated CrCL of ≥ 30 mL/min calculated by Cockcroft-Gault (using actual body weight) or serum creatinine < 2 × ULN,

   Males:

   CrCL (mL/min) = Weight (kg) × (140 - Age)/72 × serum creatinine (mg/dL)

   Females:

   CrCL (mL/min) = Weight (kg) × (140 - Age) × 0.85/72 × serum creatinine (mg/dL)
5. Meet the following laboratory parameters (Upper limit of normal (ULN) is based on institutional standards):

   1. Serum AST and ALT ≤ 3 × ULN (Higher thresholds may be allowed if hepatic dysfunction is attributable to CLL/SLL and after discussion with the Sponsor Hematology Safety Knowledge Group).
   2. Total bilirubin ≤ 1.5 × ULN, unless directly attributable to Gilbert's syndrome.
6. An ECOG (Eastern Cooperative Oncology Group) performance status performance status of 0 to 2 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
7. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).
8. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules and tablets without difficulty.

Exclusion Criteria:

1. As judged by the investigator, any evidence of past or current diseases that, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardize their safety or compliance with the protocol or would put the study at risk.
2. Clinically significant cardiovascular disease, such as symptomatic arrhythmias, congestive heart failure, or myocardial infarction, within 6 months of screening or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification. Note: Participants with controlled, asymptomatic atrial fibrillation can enroll in the study.
3. Active bleeding or history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
4. Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura.
5. History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study intervention.
6. Child-Pugh B/C liver cirrhosis.
7. History of prior or current malignancy (including but not limited to known central nervous system involvement such as by CLL/SLL, leptomeningeal disease, or spinal cord compression, known prolymphocytic leukemia or history of, or currently suspected, Richter's syndrome) that could affect compliance with the protocol or interpretation of results. Possible examples where compliance or data interpretation may not be affected could include the following, per physician discretion.

   1. Curatively treated basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin or carcinoma in situ of the cervix or carcinoma in situ of the prostate at any time prior to study.
   2. Other cancers that have been curatively treated from which the participant is disease-free for ≥ 3 years without further treatment.
8. An individual organ system dysfunction limiting the ability to receive the study intervention or any other life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the participants' safety or interfere with the absorption, distribution, metabolism, or excretion of the study interventions (eg, refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, previous significant bowel resection, or impaired resorption in the gastrointestinal tract).
9. Known history of infection with HIV or any active significant infection (eg, bacterial, viral, or fungal; including participants with positive cytomegalovirus (CMV) DNA PCR). CMV testing at screening must include serologic testing for CMV immunoglobulin G (CMV IgG), CMV immunoglobulin M (CMV IgM), and CMV DNA PCR testing. Participants must have a result for CMV DNA PCR that is negative at screening to be eligible for the study.
10. History of or ongoing confirmed progressive multifocal leukoencephalopathy (PML).
11. Serologic status reflecting active hepatitis B or C infection:

    1. Hepatitis serology will include HBsAg, anti-HBs, anti-HBc and anti-HCV. Any participant who is both anti-HBc positive and HBsAg negative will need to have a negative HBV DNA PCR result before randomization and must be willing to undergo this PCR testing during the study. Any participant who is either HBsAg positive or hepatitis B DNA PCR positive will be excluded.
    2. Participants who are hepatitis C antibody positive or inconclusive will need to have a negative HCV RNA PCR result before randomization. Those who are hepatitis C PCR positive will be excluded.
12. Any prior CLL/SLL-specific therapies, except prior rituximab if used for autoimmune cytopenias and not as anti-CLL/SLL treatment.
13. Corticosteroid use > 20 mg within 1 week before the first dose of study intervention, except as indicated for other medical conditions, such as autoimmune cytopenias, inhaled steroid for asthma, topical steroid use, or as premedication for administration of study intervention or contrast. Participants requiring steroids at daily doses > 20 mg prednisone equivalent systemic exposure daily, or those who are administered steroids for leukemia control or white blood cell count lowering, are excluded. Of note, participants may receive corticosteroids as doses > 20 mg as per institutional standards for obinutuzumab premedication prior to C1D1.
14. Prior radio- or toxin-conjugated antibody therapy.
15. Prior allogeneic stem cell or autologous transplant.
16. Known history of hypersensitivity or anaphylaxis to study intervention(s), including active product or excipient components.
17. Requires treatment with a strong cytochrome CYP3A4 inhibitor/inducer. The use of strong CYP3A inhibitors within 1 week or strong CYP3A inducers within 3 weeks of the first dose of study drug is prohibited.
18. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (other anticoagulants allowed).
19. Requires treatment with proton pump inhibitors (PPIs) (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Note: Participants receiving PPIs who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study. This criterion applies only to participants receiving acalabrutinib capsules. This PPI exclusion does not apply if the participant is receiving acalabrutinib tablets.
20. Vaccination with live vaccines 28 days prior to registration for study screening.
21. Major surgical procedure within 28 days of first dose of study intervention. Note: If a participant had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study intervention.
22. Concurrent participation in another therapeutic clinical trial. Use of investigational agents that interfere with the study intervention(s) within 28 days or 5 half-lives (whichever is longer) prior to registration for study screening.
23. Prothrombin time/INR or activated partial thromboplastin time, in the absence of lupus anticoagulant or attributed to anticoagulant (eg, direct oral anticoagulant), > 2 × ULN.
24. Currently pregnant (confirmed with positive pregnancy test) or breast feeding.
25. Women of childbearing Potential (WOCBP) unless the following criteria are met: A negative pregnancy test at least 30 days before start of study intervention, followed by immediate highly effective contraception; further pregnancy testing will be performed every cycle and as clinically indicated.
26. Fertile men or WOCBP unless the following criteria are met:

    1. Female participants (WOCBP): Willing to use highly effective contraceptive method (Pearl Index < 1 defined as failure rate of less than 1% per year when used correctly and consistently) during study intervention and for 2 days after last acalabrutinib dose, 30 days after last venetoclax dose and 18 months after last obinutuzumab dose whichever is longer.
    2. Male participants (fertile; non-sterilized): Male participants with a female partner of childbearing potential must refrain from agree to use a condom with spermicide plus an additional highly effective contraceptive method while on study treatment and 30 days after the last venetoclax dose, and 6 months after the last obinutuzumab dose, whichever is longer. These restrictions apply even if the participant had a vasectomy (condom is still needed to prevent possible direct exposure to a developing baby in case a female partner is already pregnant). Male participants must also not donate sperm during the study and for these same periods of time post-treatment.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2029-04-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Until progressive disease (PD) [assessed Up to 6.6 Years].
  To assess whether minimal residual disease (MRD)-driven finite AV treatment is NI to MRD-driven finite VO treatment with respect to PFS. PFS is defined as the time from the date of randomization until date of objective progressive disease per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 criteria as assessed by the investigator or death from any cause in the absence of progression.

SECONDARY OUTCOMES:
Rate of peripheral blood (PB) undetectable minimal residual disease (uMRD) based on a clonoSEQ^® | Screening (Days -45 through -1); Arm A (AV): Day 28 of Cycles 8, 14 and 24 and post treatment follow up visits; Arm B (VO): Day 28 of Cycles 6, 12 and 24 and post treatment follow up visits
  To assess the effect of AV treatment compared with VO treatment on uMRD at sequential time points. Rate of PB uMRD is defined as proportion of participants achieving remission based on a clonoSEQ^® assay result of < 1 CLL cell per 100,000 leukocytes (< 10 ^-5 ), after completion of 6 and 12 cycles of venetoclax (assessed at approximately 7/13 and 9/15 months for VO and AV, respectively), and at 24, 36, 48 and 60 months.
Rate of peripheral blood (PB) and Bone marrow (BM) undetectable minimal residual disease (uMRD) by flow cytometry | Cycle 14 (each Cycle length 28 days) Day 28 for Arm A (AV); Cycle 12 Day 28 for Arm B (VO) and Post treatment follow-up visits (assessed Up to 6.6 Years)
  To assess the effect of AV treatment compared with VO treatment on uMRD at sequential timepoints. Rate of PB and BM uMRD is defined as < 1 CLL cell per 10,000 leukocytes (< 10^-4) by flow cytometry, after completion of 12 cycles of venetoclax (assessed at approximately 13 and 15 months for VO and AV, respectively) and at 36 months.
Overall Survival (OS) | Date of randomization until death from any cause (Assessed Up to 6.6 Years)
  To assess the effect of AV treatment compared with VO treatment on OS. OS is defined as the time from the date of randomization until death from any cause.
Event-free Survival (EFS) | Date of randomization until first occurrence of disease progression (Assessed Up to 6.6 Years)
  To assess the effect of AV treatment compared with VO treatment on EFS. EFS is defined as the time from the date of randomization to the first occurrence of disease progression, initiation of subsequent CLL therapy, or death from any cause.
Overall Response Rate (ORR) | Date of randomization until PD (Assessed Up to 6.6 Years)
  To assess the effect of AV treatment compared with VO treatment on ORR. ORR is defined as the proportion of participants who achieve best response of Complete Response (CR), complete response with incomplete marrow recovery (Cri), nodular partial remission (nPR), or partial remission (PR) per iwCLL 2018 criteria as assessed by the investigator.
Complete Response (CR) rate | Date of randomization until PD (Assessed Up to 6.6 Years)
  To assess the effect of AV treatment compared with VO treatment on ORR. CR rate (uMRD per iwCLL guidelines 2018) after completion of 12 cycles of venetoclax.
Change from baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 scales | For AV: Cycle 1-Cycle 2, Cycle 3-Cycle 14; After End of Treatment (EoT); Post treatment follow-up For VO: Cycle 1 Day 1-21, Cycle 1 Day 22-Cycle 6, Cycle 7-Cycle 24 (Each cycle is 28 days); After EoT, Post treatment follow-up (assessed Up to 6.6 years)
  To assess symptoms, functional status and global health status/quality of life (QoL), in participants treated with AV versus VO using the EORTC QLQ-C30.
  EORTC QLQ-C30 consists of 30 items and measures symptoms, functioning, and global health status/QoL for all cancer types. Questions are grouped into 5 multi-item functional scales, 3 multi-item symptom scales, a 2-item global QoL scale, 5 single items assessing additional symptoms commonly reported by cancer participants, and 1 item on the financial impact of the disease.
  The EORTC QLQ-C30 will be scored according to the EORTC QLQ-C30 Scoring Manual. An outcome variable consisting of a score from 0 to 100 will be derived for each of the symptom scales, each of the functional scales, and the global measure of health status scale. Higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales represent greater symptom severity.
Change from baseline in EORTC QLQ-CLL17 scales | For AV: Cycle 1-Cycle 2, Cycle 3-Cycle 14; After End of Treatment (EoT); Post treatment follow-up For VO: Cycle 1 Day 1-21, Cycle 1 Day 22-Cycle 6, Cycle 7-Cycle 24 (Each cycle is 28 days); After EoT, Post treatment follow-up (assessed Up to 6.6 years)
  To assess symptoms, functional status, and global health status/QoL, participants treated with AV versus VO using the EORTC QLQ-CLL17.
  EORTC QLQ-CLL17 comprises 17 items grouped into 3 multi-item scales: 1) symptom burden, 2) physical condition/fatigue, and 3) worries/fears about health and functioning.
  The EORTC QLQ-CLL17 will be scored according to the EORTC QLQ-C30 Scoring Manual. An outcome variable consisting of a score from 0 to 100 will be derived for each of the symptom scales, each of the functional scales, and the global measure of health status scale. Higher scores on the global measure of health status and functional scales indicate better health status/function, but higher scores on symptom scales represent greater symptom severity.
Proportion of participants experiencing bruising as measured by the National Cancer Institute (NCI) Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) item for Bruising | For AV: Cycle 1-Cycle 2, Cycle 3-Cycle 14; After End of Treatment (EoT); Post treatment follow-up For VO: Cycle 1 Day 1-21, Cycle 1 Day 22-Cycle 6, Cycle 7-Cycle 24 (Each cycle is 28 days); After EoT, Post treatment follow-up (assessed Up to 6.6 years)
  To assess symptomatic toxicities patient perceived benefit-risk in participants treated with AV versus VO using the NCI PRO-CTCAE item for Bruising.
  It was designed to be used as a companion to the Common Terminology Criteria for Adverse Events (CTCAE), the standard lexicon for adverse event reporting in cancer trials. The bruising item, which has a dichotomous yes/no response option, will be included in this study to capture patient-reported bruising.
Proportion of participants reporting each response option of the Patient Global Impression of Benefit-Risk (PGI-BR) | For AV: Cycle 1-Cycle 2, Cycle 3-Cycle 14 (Each cycle is 28 days); and End of treatment, E/D, disease progression, and post-treatment follow-up visits (assessed up to 6.6 years)
  To assess patient perceived benefit-risk of treatment in participants treated with AV versus VO using the PGI-BR.
  PGI-BR consists of 4 study medication-related questions, one each on efficacy, side effects, convenience of use, and overall benefit-risk. Each item is scored separately, with the final item providing a single metric of a participant's overall benefit-risk assessment.
  The response from each question will be semi-quantitative. Each question ranges from Very (negative, Somewhat [negative]), Neutral, Somewhat [positive], Very [positive].
Number of participants with adverse events (AEs) | From screening (Days -45 through -1) until survival follow-up (Up to 6.6 years)
  To assess the safety and tolerability of AV treatment versus VO treatment in participants with previously untreated CLL/SLL.

CONTACTS AND LOCATIONS:
Locations (37):
- United States (18):
  - Research Site, Tucson, Arizona
  - Research Site, La Jolla, California
  - Research Site, Longmont, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
- Australia (4):
  - Research Site, Clayton
  - Research Site, Geelong
  - Research Site, Nedlands
  - Research Site, Waratah
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Ostrava - Poruba
  - Research Site, Pilsen
- France (2):
  - Research Site, Montpellier
  - Research Site, Tours
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Debrecen
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lódz
  - Research Site, Lublin
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ryan CE, Davids MS, Hermann R, Shahkarami M, Biondo J, Abhyankar S, Alhasani H, Sharman JP, Mato AR, Roeker LE. MAJIC: a phase III trial of acalabrutinib + venetoclax versus venetoclax + obinutuzumab in previously untreated chronic lymphocytic leukemia or small lymphocytic lymphoma. Future Oncol. 2022 Oct;18(33):3689-3699. doi: 10.2217/fon-2022-0456. Epub 2022 Sep 14. PMID 36102212